CLINICAL TRIAL: NCT01084486
Title: Effect of Treatment With Insulin Sensitizer on Arterial Properties, Metabolic Parameters and Liver Function in Patients With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Other Study IDs: WolfsonMC-2007-9
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: nonalcoholic fatty liver disease; Pulse wave velocity; augmentation index; metformin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Metformin

ARMS (1):
- Metformin, Adiponectine, Arterial Compliance (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Abstract

Background: Insulin resistance has an important role in the development of nonalcoholic fatty liver disease (NAFLD) and is involved in both pathological processes: hepatic steatosis and atherosclerosis. Therefore, treatment of NAFLD with insulin sensitizers is likely to have a favorable effect towards hepatic steatosis and cardiovascular outcomes.

Objectives: The present study investigated the effect of metformin on arterial properties, metabolic parameters and liver function in patients with NAFLD. Methods In randomized, placebo controlled study, 63 patients with NAFLD were assigned to one of two groups: Group 1 received daily metformin; Group 2 received placebo. Pulse wave velocity (PWV) and augmentation index (AI) were performed using SphygmoCor (version 7.1, AtCor Medical, Sydney, Australia) at baseline and at the end of 4-month treatment period.. Metabolic measures and serum adiponectin levels were determined.

ELIGIBILITY:
Inclusion Criteria:

* In a single-center study, 63 patients (32 males and 31 females) diagnosed with nonalcoholic fatty liver disease were recruited from the outpatient clinic and evaluated for the study.

Exclusion Criteria:

* Patients with history of unstable angina, MI, CVA or major surgery within the six months preceding entrance to the study.
* Patients with unbalanced endocrine disease or any disease that might affect absorption of medications.
* Patients with plasma creatinine > 1.5 mg/dl, and electrolyte abnormalities.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel

REFERENCES:
- [Derived] Sofer E, Shargorodsky M. Effect of metformin treatment on circulating osteoprotegerin in patients with nonalcoholic fatty liver disease. Hepatol Int. 2016 Jan;10(1):169-74. doi: 10.1007/s12072-015-9649-6. Epub 2015 Jul 22. PMID 26198758
- [Derived] Shargorodsky M, Omelchenko E, Matas Z, Boaz M, Gavish D. Relation between augmentation index and adiponectin during one-year metformin treatment for nonalcoholic steatohepatosis: effects beyond glucose lowering? Cardiovasc Diabetol. 2012 Jun 7;11:61. doi: 10.1186/1475-2840-11-61. PMID 22676459
- [Derived] Sofer E, Boaz M, Matas Z, Mashavi M, Shargorodsky M. Treatment with insulin sensitizer metformin improves arterial properties, metabolic parameters, and liver function in patients with nonalcoholic fatty liver disease: a randomized, placebo-controlled trial. Metabolism. 2011 Sep;60(9):1278-84. doi: 10.1016/j.metabol.2011.01.011. Epub 2011 Mar 15. PMID 21411114